CLINICAL TRIAL: NCT03050866
Title: A Single Arm Phase 2 Multicenter Study Determining the Response to Cabazitaxel in Metastatic Prostate Cancer (mCRPC) Patients With AR-V7 Positive Circulating Tumor Cells (CTCs)
Brief Title: Cabazitaxel in mCRPC Patients With AR-V7 Positive Circulating Tumor Cells (CTCs)
Acronym: CABA-V7
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, M.P.J.K. Lolkema, Dr., Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL58639.056.16
Record Dates: First submitted 2017-02-07; First posted 2017-02-13 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Circulating Tumor Cell; Metastatic Prostate Cancer
Keywords: Androgen Receptor; AR-V7; Predictive Factor
MeSH Terms: conditions — Neoplastic Cells, Circulating; Prostatic Neoplasms; Bulbo-Spinal Atrophy, X-Linked | interventions — cabazitaxel; Histamine Antagonists; Adrenal Cortex Hormones; Histamine H2 Antagonists; Antiemetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Other): Treatment intervention with Cabazitaxel with premedication as necessary (antihistamine, corticosteroid, H2 antagonist, antiemetic prophylaxis)
  Interventions: Drug: Cabazitaxel; Other: Antihistamine; Other: Corticosteroid; Other: H2 antagonist; Other: Antiemetic

INTERVENTIONS:
Drug: Cabazitaxel — 25mg/m2 q3w
  Other Names: Jevtana
Other: Antihistamine — As intravenous premedication (dexchlorpheniramine 5 mg, diphenhydramine 25 mg, or equivalent)
Other: Corticosteroid — As intravenous premedication (dexamethasone 8 mg or equivalent)
Other: H2 antagonist — As intravenous premedication (ranitidine or equivalent)
  Other Names: histamine H2 receptors blockers
Other: Antiemetic — Antiemetic prophylaxis is recommended and can be given orally or intravenously if necessary

SUMMARY:
After failure on docetaxel, which has been the standard first line therapy for patients with metastatic castration-resistant prostate cancer (mCRPC), several treatment options are currently available.

In retrospective studies, resistance has been described to two of the treatment options, enzalutamide and abiraterone, when a splice variant of the Androgen Receptor (AR-V7) is present on circulating tumor cells (CTCs). The investigators hypothesize that patients with AR-V7 positive CTCs do have a meaningful response to cabazitaxel.

DETAILED DESCRIPTION:
After failure on docetaxel, which has been the standard first line therapy for patients with metastatic castration-resistant prostate cancer (mCRPC), several treatment options are currently available.

Two of the treatment options are directed against the androgen receptor (AR), enzalutamide and abiraterone. A third option is cabazitaxel, a next generation taxane. No head-to-head comparisons have been done for these three therapies in second-line mCRPC and as of yet, the optimal choice is unknown.

Resistance to the AR-targeted therapies is at least in part a consequence of signaling through constitutively active AR splice variants (AR-Vs). Because AR splice variants only occur after conversion to a castration-resistant tumor, and can be acquired during systemic therapy for mCRPC, analysis of the castration-naïve primary tumor is not informative in the setting of second-line treatment of mCRPC.

Circulating tumor cells (CTCs) can be analyzed repetitively and in real-time. Recently, AR-V7 messenger ribonucleid acid (mRNA) expression in CTCs was shown to be associated with lack of response to AR-targeted therapy (reference 1). AR-V7 mRNA expression does not seem to hinder response to cabazitaxel in our retrospective pilot study (reference 2) nor in two recently published retrospective studies (reference 3 and reference 4).

Therefore we hypothesize that the mRNA expression of AR-V7 in CTCs assessed before start of second-line treatment for mCRPC does not affect prostate-specific antigen (PSA) response to cabazitaxel in patients who have progressed to docetaxel.

Patients who are eligible to undergo second or third line treatment will be asked to undergo prescreening consisting of a CTC count and, in case ≥3 CTCs are detected, AR V7 determination. Patients with ≥3 CTCs with AR-V7 expression will be asked to sign a second informed consent to enter the treatment study. In this study they will receive Cabazitaxel 25 mg/m² every 3 weeks plus prednisone 10 mg daily, and undergo repeated blood sampling for biomarker sample collection.

During the prescreening in all patients, 2 x 10 mL blood will be drawn for enumeration and isolation of CTCs. All patients with ≥3 CTCs with AR-V7 expression will be asked to sign consent for the treatment study.

All patients included in the treatment study will be administrated cabazitaxel intravenously at a dose of 25 mg/m², during a one-hour infusion every 3 weeks, as well as continuous treatment with prednisone 5 mg orally twice daily, or 10 mg once daily. In the treatment study patients, an additional 2 x 10 mL blood will be drawn after the third cycle of treatment for CTC enumeration and isolation. An additional 10 mL blood will be drawn for storage of plasma at baseline and before start of every cycle (i.e., every 3 weeks) for analysis of cell-free DNA (cfDNA). Moreover, 4 x 5 mL blood (baseline; end of infusion, 2 and 6 hours after end of the first cabazitaxel infusion) will be drawn for pharmacokinetic studies, in order to explore a cabazitaxel exposure effect relation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features.
* Continued androgen deprivation therapy either by luteinizing hormone-releasing hormone (LHRH) agonists/antagonists or orchiectomy.
* Serum testosterone <50 ng/mL (1.7 nmol/L) within 21 days before prescreening.
* Age ≥18 years
* Received prior docetaxel, and experienced disease progression during or after treatment with docetaxel.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (appendix A)
* Written informed consent according to ICH-GCP (International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use - Good Clinical Practice) before study treatment and any study specific procedures

Exclusion Criteria:

* Geographical, psychological or other non-medical conditions interfering with follow-up
* Uncontrolled severe illness or medical condition (including uncontrolled diabetes mellitus or active systemic or local bacterial, viral, fungal - or yeast infection)
* Symptomatic central nervous system (CNS) metastases or history of psychiatric disorder that would prohibit the understanding and giving of informed consent.
* Chemotherapy or immunotherapy (other than LHRH analogues) within the last 4 weeks before study inclusion.
* Prior treatment with cabazitaxel
* Treatment with both abiraterone and enzalutamide in the post-docetaxel setting
* Radiotherapy to 40% or more of the bone marrow
* Known hypersensitivity to corticosteroids
* History of severe hypersensitivity reaction (≥grade 3) to docetaxel
* History of severe hypersensitivity reaction (≥grade 3) to polysorbate 80 containing drugs
* Concurrent or planned treatment with strong inhibitors or strong inducers of cytochrome P450 3A4/5 (a one week wash-out period is necessary for patients who are already on these treatments)
* Concomitant vaccination with yellow fever vaccine
* Abnormal liver functions
* Abnormal hematological blood counts

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2017-02-21 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-08-19 (Estimated)

PRIMARY OUTCOMES:
PSA response | 12 weeks after start of treatment
  The primary endpoint is PSA response, defined as a ≥50% PSA decline from baseline during therapy.

SECONDARY OUTCOMES:
CTC response | 9-12 weeks after start of treatment
  CTC response defined as a decrease from ≥5 CTCs per 7.5 mL blood at baseline to <5 CTCs per 7.5 mL blood
PSA change | 12 weeks after start of treatment
  PSA change from baseline at 12 weeks defined as the percent change in PSA from baseline at 12 weeks, according to PCWG2 criteria
PSA decrease | PSA will be assessed at baseline, every 3 weeks during study treatment (before every cycle), and in case of study treatment discontinuation without progression every 3 months until progression, death, whichever comes first
  Maximum PSA decrease defined according to PCWG2 criteria
Progression free survival | Until end of study, which is anticipated to be 4 years after inclusion of first patient. If progression is not observed during the study, data on PFS will be censored
  Progression-free survival (PFS) defined as time from prescreening to the date of the first documentation of disease progression (PCWG2)
Overall survival | Until end of study, which is anticipated to be 4 years after inclusion of first patient. If death is not observed during the study, data on OS will be censored at the date patient is known to be alive or at the cut-off date, whichever comes first
  Overall survival (OS) calculated from the date of prescreening to death due to any cause
Adverse Events | Until 30 days after end of treatment, Cabazitaxel treatment will consist of a maximum 10 cycles Cabazitaxel (given once every 3 weeks if there are no delays)
  Grade 3-4 adverse events (AEs) and serious adverse events (SAEs) during cabazitaxel according to CTCAE v4.03 in second and third-line treatment
Cumulative dose Cabazitaxel | Until last day of administration of study medication (Cabazitaxel), Cabazitaxel treatment will consist of a maximum 10 cycles Cabazitaxel (given once every 3 weeks if there are no delays)
  Cumulative administered dose of cabazitaxel in second and third-line treatment
Splice variants | Splice variant will be compared before and after cabazitaxel treatment in AR-V7 positive patients, as well as before start of enzalutamide or abiraterone and after disease progression to this treatment.
  AR-V7 mRNA expression as well as mRNA expression of other splice variants in CTCs indicated as absent (-) or present (+)
Total systemic exposure | After infusion of first cycle of study treatment (Cabazitaxel)
  Cabazitaxel concentration in the blood and total systemic exposure to cabazitaxel, measured by the calculated area under the curve (AUC)
Value ctDNA quantification | Until end of study, which is anticipated to be 4 years after inclusion of first patient
  To explore the value of ctDNA quantification during cabazitaxel treatment to predict tumor progression

CONTACTS AND LOCATIONS:
Locations (9):
- Netherlands (9):
  - Reinier de Graaf Groep, Delft
  - Admiraal de Ruyter Ziekenhuis, Flushing
  - Groene Hart Ziekenhuis, Gouda
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Erasmus MC, Rotterdam
  - Franciscus Gasthuis en Vlietland, Rotterdam
  - Maasstad Ziekenhuis, Rotterdam
  - Medisch Centrum Haaglanden, The Hague
  - Tweesteden Ziekenhuid, Tilburg

IPD SHARING:
Plan to Share IPD: Undecided
Information can be shared by importing it into another databases